CLINICAL TRIAL: NCT06830629
Title: An Open-Label Phase 2 Study to Evaluate the Safety, Tolerability, and Effect on Albuminuria of MZE829 in Adults With Proteinuric Chronic Kidney Disease and the APOL1 High Risk Genotype
Brief Title: A Phase 2 Study of MZE829 in Adults With APOL1 Kidney Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Maze Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MZE829-201
Record Dates: First submitted 2025-02-07; First posted 2025-02-17 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Proteinuric Kidney Disease
Keywords: APOL1-mediated kidney disease (AMKD); APOL1 kidney disease (AKD)

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MZE829 (Experimental): Cohort 1: Chronic kidney disease with concurrent diabetes
  Cohort 2: Chronic kidney disease without concurrent diabetes
  Interventions: Drug: MZE829

INTERVENTIONS:
Drug: MZE829 — Capsules for oral administration

SUMMARY:
This is purpose of this study is to evaluate the safety, tolerability, and effect on Albuminuria of MZE829 in Adults with APOL1 Kidney Disease

DETAILED DESCRIPTION:
An open-label Phase 2 study is designed to evaluate the safety, tolerability, and effect on Albuminuria of MZE829 in Adults with Proteinuric Chronic Kidney Disease and the APOL1 High Risk Genotype.

ELIGIBILITY:
Key Inclusion Criteria:

* APOL1 high risk genotype of G1/G1, G2/G2, or G1/G2
* Chronic kidney disease with persistent albuminuria

Key Exclusion Criteria:

* Organ or bone marrow transplantation
* History of cancer within past 2 years, excepted for treated non-melanoma skin cancer, stage 0 cervical cancer, or stage 1 prostate cancer
* Conditions that may alter drug absorption, e.g., history of bariatric surgery
* Type I diabetes
* Pregnant or currently nursing

Other inclusion/exclusion criteria defined in protocol apply.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by incidence of adverse events (AEs) | Day 1 to Week 12

SECONDARY OUTCOMES:
Percent participants with ≥30% reduction from baseline in UACR at Week 12 | Day 1 to Week 12
Geometric mean plasma drug concentrations | Day 1 to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Maze Therapeutics
Locations (67):
- United States (61):
  - Research Site, Decatur, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Montgomery, Alabama
  - Research Site, Granada Hills, California
  - Research Site, Bloomfield, Connecticut
  - Research Site, Atlantis, Florida
  - Research Site, Brandon, Florida
  - Research Site, Brooksville, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Orlando, Florida
  - Research Site, College Park, Georgia
  - Research Site, Cordele, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Riverdale, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Kansas City, Kansas
  - Research Site, Bowling Green, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Arnold, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Lutherville, Maryland
  - Research Site, Oxon Hill, Maryland
  - Research Site, Dearborn, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Saint Joseph, Michigan
  - Research Site, Shelby, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Fayette, Mississippi
  - Research Site, Ridgeland, Mississippi
  - Research Site, Tupelo, Mississippi
  - Research Site, City of Saint Peters, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Laurelton, New York
  - Research Site, Maspeth, New York
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Fayetteville, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Shelby, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Ardmore, Oklahoma
  - Research Site, Upland, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Greenville, Texas
  - Research Site, Houston, Texas
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Shenandoah, Texas
  - Research Site, Sherman, Texas
  - Research Site, Hampton, Virginia
  - Research Site, Norfolk, Virginia
- France (4):
  - Research Site, Créteil
  - Research Site, Lyon
  - Research Site, Paris
  - Research Site, Saint-Ouen
- United Kingdom (2):
  - Research Site, Leicester
  - Research Site, London

IPD SHARING:
Plan to Share IPD: No